CLINICAL TRIAL: NCT04571658
Title: Implementing Precision Medicine for Glomerular Diseases in the Nephrotic Syndrome Study Network (NEPTUNE)
Brief Title: NEPTUNE Match Study
Acronym: NEPTUNE Match
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Matthias Kretzler, Internal Medicine Professor, University of Michigan
Other Study IDs: HUM00158219-Sub; U54DK083912 (NIH)
Record Dates: First submitted 2020-09-08; First posted 2020-10-01 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Nephrotic Syndrome in Children; Focal Segmental Glomerulosclerosis; Minimal Change Disease; Minimal Change Nephrotic Syndrome; Membranous Nephropathy; FSGS; MCD; MCD - Minimal Change Disease; Alport Syndrome
Keywords: Nephrotic Syndrome; NEPTUNE; Match; Clinical Trial Match
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Nephrosis, Lipoid; Glomerulonephritis, Membranous; Macular dystrophy, corneal type 1; Nephritis, Hereditary; Nephrotic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and Urine as part of the NEPTUNE study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NEPTUNE Match Participants: Approximately 375 participants will be consented from the NEPTUNE observational study with age and demographic groups representing the patient population in the NEPTUNE study site geographical areas.
  NEPTUNE observational cohort eligibility includes: participants in NEPTUNE observational cohort A are of any age and have a biopsy-confirmed diagnosis of Focal Segmental Glomerulosclerosis (FSGS), Minimal Change Disease (MCD), or Membranous Nephropathy (MN). Participants in NEPTUNE observational cohort B have documented NS based on proteinuria, serum albumin, and/or edema with age of onset less than 19 years.
  Interventions: Other: Communication

INTERVENTIONS:
Other: Communication — The NEPTUNE Match study includes an interdisciplinary Communication Team that will translate findings from the Molecular Nephrology Board (MNB) to inform patients of the matching assessment with ongoing clinical trials. This team has considerable experience with conveying complex biomedical research information to patients and families and includes experts in precision nephrology, nephrology patient [adult and pediatric] communication, and health education.

SUMMARY:
NEPTUNE Match is an additional opportunity offered to NEPTUNE study participants to prospectively recruit and communicate patient-specific clinical trial matching with kidney patients and their physician investigators.

DETAILED DESCRIPTION:
This is a prospective, open-label study testing the ability to effectively communicate patient-specific clinical trial matching with kidney patients and clinician investigators. The study consists of four components:

1. Recruitment of participants from the NEPTUNE observational cohort study
2. Generation of participant profile-trial match assessment using data from the NEPTUNE observational study and profiling units by the NEPTUNE Molecular Nephrology Board
3. Establishing and testing a framework to communicate disease-trial drug mechanism matching with investigators and patients
4. Retrospective comparison of kidney health outcomes in subjects enrolled in trials that aligned with their match vs. trial subjects with mis-aligned or unknown match alignment.

ELIGIBILITY:
Inclusion Criteria:

1. Consented and eligible participants in the biopsied or non-biopsied cohorts of the NEPTUNE observational study
2. Must be potentially eligible for the NEPTUNE Match partnering trials (e.g. if no trial is enrolling a participant under age 6, those under 6 are not eligible).

   Note: NEPTUNE Match partnering trials and associated eligibility criteria are expected to be dynamic and change as trial protocols are developed, activated, and amended.
3. Regular nephrology healthcare provided at a NEPTUNE study site.
4. Willing and able to consent, and as appropriate assent, to participate in NEPTUNE Match

Exclusion Criteria:

Currently non-NEPTUNE observational study participants are not eligible to be matched to a clinical trial using these biomarker assessments.

Exclusion Criteria:

1. Non-English or non-Spanish speaking

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from the NEPTUNE observational cohort within NEPTUNE clinical sites by trained and experienced study teams. Enrollment into the NEPTUNE observational cohorts and NEPTUNE Match will be ongoing, parallel activities. However participants must be confirmed eligible for inclusion in the NEPTUNE observational study before they are enrolled into NEPTUNE Match. If a NEPTUNE observational study participant previously completed the final NEPTUNE visit, they may undergo a re-enrollment visit in the NEPTUNE III observational study as NEPTUNE III will be open to prevalent patients.
Sampling Method: Non-Probability Sample
Enrollment: 375 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Matched participants with at least one clinical trial receive a MNB assessment | 0-4 weeks
  Proportion of NEPTUNE Match participants with at least one matching clinical trial, defined as receiving a Molecular Nephrology Board (MNB) assessment that provides a match to at least one targeted therapy in an ongoing clinical trial
Efficacy of communication methods at time of communication visit, measured by Teach Back 1 summary score | 12 weeks
  Key findings from MNB trial matching analyses and deliberations will be conveyed to study participants using a NEPTUNE Match Report that summarizes the findings. The report indicates the strength of matching to ongoing clinical trials and the uncertainty and research origins of the information. A sample Match Report can be found in Appendix C. The report will not contain individual data elements reviewed by the MNB. The creation of NEPTUNE Match Reports will follow health education principles including matching of content to patients' informational needs and health literacy levels, use of visual aids to clarify meaning of information, and avoidance of information overload of the participant.
Kidney health endpoints that are specific to each individual trial | 0-60 months
  The analytic integration supporting the Molecular Nephrology Board (MNB) case review will be initiated and will occur. The MNB will conduct the discussion and generate the integrated data summary and case report inclusive of clinical trial matching by webinar. Input from the MNB will be used to generate a final version of the participant NEPTUNE Match Report. This is a longitudinal outcome that will be assessed at the end of the study relative to endpoints specific to matched clinical trials, assessing the superiority of stratification (matching or alignment of patient molecular profiles to targeted therapies in clinical trials) to non-stratification.

SECONDARY OUTCOMES:
Efficacy of communication methods at follow up, measured by Teach Back of key concepts | 14-18 weeks
  3 defined teachback concepts will be scored to indicate the participant's understanding of strength of matching.
Psychological distress measured by the STAI assessment | 14-18 weeks
  State Trait Anxiety Inventory (mini-STAI) scale will be used to assess a participant's psychological distress around their participation in NEPTUNE Match at the consent visit and the follow up visit.
Psychological distress measured by the FACToR-NEPTUNE assessment | 14-18 weeks
  FACToR-NEPTUNE is a measure that has been modified from the Feelings About genomiC Testing Results (FACToR). FACToR-12 is used to assess the psychosocial impact of returning genomic findings to patients in research and clinical practice. In the FACToR-NEPTUNE assessment the measure will assess the psychosocial impact after receiving the NEPTUNE Match Report.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Kretzler, MD, Principal Investigator — University of Michigan; Debbie GIpson, MD, MS, Study Director — University of Michigan
Locations (16):
- United States (16):
  - Emory University Hospital - Children's Hospital of Atlanta, Atlanta, Georgia
  - John H. Stroger, Jr., Hospital of Cook County, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins Medicine, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - Northwell/Cohen's Children's Hospital, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charlotte, South Carolina
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Providence Sacred Heart Medical Center, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gadegbeku CA, Gipson DS, Holzman LB, Ojo AO, Song PX, Barisoni L, Sampson MG, Kopp JB, Lemley KV, Nelson PJ, Lienczewski CC, Adler SG, Appel GB, Cattran DC, Choi MJ, Contreras G, Dell KM, Fervenza FC, Gibson KL, Greenbaum LA, Hernandez JD, Hewitt SM, Hingorani SR, Hladunewich M, Hogan MC, Hogan SL, Kaskel FJ, Lieske JC, Meyers KE, Nachman PH, Nast CC, Neu AM, Reich HN, Sedor JR, Sethna CB, Trachtman H, Tuttle KR, Zhdanova O, Zilleruelo GE, Kretzler M. Design of the Nephrotic Syndrome Study Network (NEPTUNE) to evaluate primary glomerular nephropathy by a multidisciplinary approach. Kidney Int. 2013 Apr;83(4):749-56. doi: 10.1038/ki.2012.428. Epub 2013 Jan 16. PMID 23325076
- [Background] Tao J, Mariani L, Eddy S, Maecker H, Kambham N, Mehta K, Hartman J, Wang W, Kretzler M, Lafayette RA. JAK-STAT signaling is activated in the kidney and peripheral blood cells of patients with focal segmental glomerulosclerosis. Kidney Int. 2018 Oct;94(4):795-808. doi: 10.1016/j.kint.2018.05.022. Epub 2018 Aug 6. PMID 30093081
- [Background] Ha Dinh TT, Bonner A, Clark R, Ramsbotham J, Hines S. The effectiveness of the teach-back method on adherence and self-management in health education for people with chronic disease: a systematic review. JBI Database System Rev Implement Rep. 2016 Jan;14(1):210-47. doi: 10.11124/jbisrir-2016-2296. PMID 26878928
- [Background] Marteau TM, Bekker H. The development of a six-item short-form of the state scale of the Spielberger State-Trait Anxiety Inventory (STAI). Br J Clin Psychol. 1992 Sep;31(3):301-6. doi: 10.1111/j.2044-8260.1992.tb00997.x. PMID 1393159
- [Background] Tluczek A, Henriques JB, Brown RL. Support for the reliability and validity of a six-item state anxiety scale derived from the State-Trait Anxiety Inventory. J Nurs Meas. 2009;17(1):19-28. doi: 10.1891/1061-3749.17.1.19. PMID 19902657
- See also: Redefining Nephrotic Syndrome in Molecular Terms: Outcome-associated molecular clusters and patient stratification with noninvasive surrogate biomarkers — http://dx.doi.org/10.1101/427880
- See also: Teachback — http://www.ahrq.gov/patient-safety/reports/engage/interventions/teachback.html
- See also: Are physicians and patients in agreement? Exploring dyadic concordance — http://dx.doi.org/10.1016/j.jpainsymman.2006.11.009
- See also: Patients' memory for medical information — http://dx.doi.org/10.1258
- See also: Patient information recall in a rheumatology clinic — http://dx.doi.org/10.1093/rheumatology/18.1.18
- See also: Inflammatory and JAK-STAT Pathways as Shared Molecular Targets for ANCA-Associated Vasculitis and Nephrotic Syndrome — http://doi.org/10.1101/427898